CLINICAL TRIAL: NCT01113710
Title: Non-Interventional Study (NIS) in Patients With Restless Legs Syndrome (RLS) to Assess the Effectiveness and Safety of Neupro® in Daily Practise
Brief Title: Non-interventional Study (NIS) in Patients With Restless Legs Syndrome in Daily Practise
Acronym: RLS-Practise
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SP0948
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-08

CONDITIONS: Idiopathic Restless Legs Syndrome
Keywords: Rotigotine; Neupro®; Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neupro®: Routine treatment in accordance with the local marketing authorization for Neupro® in RLS
  Interventions: Drug: Neupro®

INTERVENTIONS:
Drug: Neupro® — Neupro® is the exposure/intervention of interest in this non-interventional study.

SUMMARY:
This non-interventional observational study is designed to gain data for Neupro® in restless legs syndrome (RLS) under real life conditions in line with the summary of product characteristics (SmPC) related to effectiveness, tolerability and switching practice from other dopaminergic drugs as well as titration schemes.

DETAILED DESCRIPTION:
There is a total of 64 subjects recorded as having discontinued due to Adverse Events. Documentation of Visit 2 and Visit 3, where the reason for discontinuation was documented, was not available for all subjects. From the documentation on the Adverse Events page in the Case Report Form, it is known that 100 subjects discontinued due to Adverse Events.

The Last Observation Carried Forward (LOCF) method was utilized for all outcomes.

ELIGIBILITY:
Inclusion Criteria:

* It was recommended that the patient's treatment was in accordance with the local marketing authorization (MA) for Neupro®
* The patient must have a diagnosis of moderate to severe idiopathic RLS
* The patient is considered reliable and capable of adhering to the visit schedule or medication administration according to the judgment of the investigator
* The decision to prescribe the drug has been made by the physician independently of his/her decision to include the patient in the study
* Subject is informed and given ample time and opportunity to think about his/her participation in the study and has given written informed data consent

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Magnetic resonance imaging or cardioversion (see SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of moderate to severe idiopathic RLS treated with Neupro® in routine daily practice.
Sampling Method: Non-Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (80):
- Germany (80):
  - Abensburg
  - Altenholz
  - Alzenau in Unterfranken
  - Anklam
  - Aschaffenburg
  - Bad Neustadt an der Saale
  - Berlin
  - Bielefeld
  - Bischofswerda
  - Bochum
  - Bonn
  - Böblingen
  - Bremen
  - Cologne
  - Cottbus
  - Delbrück
  - Dippoldiswalde
  - Dortmund-Kirchhörde
  - Dresden
  - Düren
  - Ellwangen
  - Erbach im Odenwald
  - Freiburg im Breisgau
  - Fulda
  - Gelsenkirchen
  - Gera
  - Gladenbach
  - Göttingen
  - Greifswald
  - Gütersloh
  - Halle
  - Heidenheim
  - Ilmenau
  - Jülich
  - Karlsruhe
  - Karlstadt am Main
  - Kassel
  - Kaufbeuren
  - Kleve
  - Königsbrück
  - Leipzig
  - Lemgo
  - Leun-Biskirchen
  - Lippstadt
  - Lohr a. Main
  - Ludwigsfelde
  - Malchin
  - Mannheim
  - Marburg
  - Marburg-Cappel
  - München
  - Neuburg an der Donau
  - Neusäß
  - Oberursel
  - Oelde
  - Osnabrück
  - Osterode am Harz
  - Paderborn
  - Potsdam
  - Remscheid
  - Rheda-Wiedenbrück
  - Rostock
  - Schriesheim
  - Schwalmstadt-Treysa
  - Schwäbisch Gmünd
  - Schwedt
  - Schwerin
  - Senftenberg
  - Soest
  - Stadtroda
  - Stralsund
  - Stuttgart
  - Teupitz
  - Ulm
  - Westerstede
  - Wiesbaden
  - Wismar
  - Wolfsburg
  - Zschadrass
  - Zwickau

REFERENCES:
- [Derived] Stiasny-Kolster K, Berg D, Hofmann WE, Berkels R, Grieger F, Lauterbach T, Schollmayer E, Bachmann CG. Effectiveness and tolerability of rotigotine transdermal patch for the treatment of restless legs syndrome in a routine clinical practice setting in Germany. Sleep Med. 2013 Jun;14(6):475-81. doi: 10.1016/j.sleep.2013.02.013. Epub 2013 May 11. PMID 23668924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started in May 2010 with subjects from Germany. The study completed in July 2011. The Full Analysis Set is used for study outcome measures.
  The Enrolled Set is reflected in the Participant Flow and Study Demographics. Age demographic information is missing for 1 subject and gender information is missing for 5 subjects.
Pre-assignment Details: The Participant Flow contains single and multiple reasons for "Other" subject discontinuation. Therefore, individual "Other" reasons are listed below:
  Augmentation: 7
  Problems with adhesiveness of patch: 6
  Pruritus: 1
  Tiredness: 1
  Less effective than previous medication: 1
  Application site reactions: 2
  Neurotic: 1
Period: Overall Study
Arm/Group | Neupro®
Started | 687 (See Additional Study Description for further information regarding withdrawal due to Adverse Event.)
Completed | 418 (Discontinued reasons for "Other" are listed in the Participant Flow.)
Not Completed | 269
Not completed — Adverse Event | 64
Not completed — Lack of Efficacy | 41
Not completed — No Information Available | 40
Not completed — Withdrawal by Subject | 28
Not completed — Lost to Follow-up | 20
Not completed — Lack of Efficacy/Withdrawal by Subject | 13
Not completed — Withdrawal by Subject/Adverse Event | 11
Not completed — Lack of Patient's Compliance | 8
Not completed — Other | 7
Not completed — Adverse Event/Other | 5
Not completed — Patient's Compliance/Lost to Follow up | 5
Not completed — Lack of Efficacy/Other | 4
Not completed — Patient Compliance/Withdrawal by Subject | 4
Not completed — Lack of Efficacy/Adverse Event | 3
Not completed — Efficacy/Subject Withdrawal/AE | 2
Not completed — Compliance/Lost to Follow up/Pt Withdraw | 2
Not completed — Lost to Follow up/Withdrawal by Subject | 2
Not completed — Efficacy/Withdrawal by Subject/Other | 1
Not completed — Compliance/Efficacy/Adverse Event | 1
Not completed — Compliance/Efficacy/AE/Other | 1
Not completed — Compliance/Efficacy/Subject Withdrawal | 1
Not completed — Compliance/Lost to Follow up/Efficacy/AE | 1
Not completed — Lack of Patient's Compliance/Other | 1
Not completed — Compliance/Subject Withdrawal/AE | 1
Not completed — Subject Did Not Receive Neupro | 3

BASELINE CHARACTERISTICS:
Arm/Group | Neupro®
Number analyzed (Participants) | 687
Age Continuous [Mean (Standard Deviation); unit: years] | 65.6 (12.6)
Age, Customized [Number; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 278
  >=65 years | 408
  Missing | 1
Sex/Gender, Customized [Number; unit: Participants]
  Female | 494
  Male | 188
  Missing | 5
Region of Enrollment [Number; unit: participants]
  Germany | 687

OUTCOME MEASURES:

1. Primary Outcome: Severity of Restless Legs Syndrome (RLS) at Bedtime
Description: Severity of RLS at bedtime measured as change from baseline to end of observation period (Item 2 RLS-6 scale).
  The Last Observation Carried Forward (LOCF) method was utilized for all outcomes.
  The RLS-6 scale is an 11-point scale (from 0 = not present/completely satisfied to 10 = very severe/completely dissatisfied) to establish an individual severity profile at various day and night times (at bedtime; during the night; during the day when the patients are resting, or during the day when the patients are involved in daily activities).
Time Frame: From Baseline to end of Observation Period (3 months).
Population: Of the 564 subjects in the Full Analysis Set (FAS), 564 are included in this analysis.
  The FAS consists of all patients receiving treatment with Rotigotine at least once & for whom valid scores for item 2 & item 3 of the RLS-6 scale at baseline & at least one valid post baseline score for both item 2 & item 3 of the RLS-6 scale is documented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro®
Number analyzed (Participants) | 564
units on a scale
  Change from Baseline to End of Observation Period | -2.2 (3.6)
  Observed Value at Baseline Visit | 5.2 (3.2)

2. Primary Outcome: Severity of Restless Legs Syndrome (RLS) During the Night
Description: Severity of RLS during the night measured as change from baseline to end of observation period (Item 3 RLS-6 scale).
  The Last Observation Carried Forward (LOCF) method was utilized for all outcomes.
  The RLS-6 scale is an 11-point scale (from 0 = not present/completely satisfied to 10 = very severe/completely dissatisfied) to establish an individual severity profile at various day and night times (at bedtime; during the night; during the day when the patients are resting, or during the day when the patients are involved in daily activities).
Time Frame: From Baseline to end of Observation Period (3 months).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro®
Number analyzed (Participants) | 564
units on a scale
  Change from Baseline to End of Observation Period | -2.5 (3.4)
  Observed Value at Baseline Visit | 5.5 (2.9)

3. Secondary Outcome: Satisfaction With Sleep
Description: Satisfaction with sleep measured as change from baseline to end of observation period (Item 1 RLS-6 scale).
  The Last Observation Carried Forward (LOCF) method was utilized for all outcomes.
  The RLS-6 scale is an 11-point scale (from 0 = not present/completely satisfied to 10 = very severe/completely dissatisfied) to establish an individual severity profile at various day and night times (at bedtime; during the night; during the day when the patients are resting, or during the day when the patients are involved in daily activities).
Time Frame: From Baseline to end of Observation Period (3 months).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro®
Number analyzed (Participants) | 564
units on a scale
  Change from Baseline to End of Observation Period | -2.4 (3.5)
  Observed Value at Baseline Visit | 6.4 (2.7)

4. Secondary Outcome: Severity of Restless Legs Syndrome (RLS) at Daytime at Rest
Description: Severity of RLS at daytime at rest measured as change from baseline to end of observation period (Item 4 RLS-6 scale).
  The Last Observation Carried Forward (LOCF) method was utilized for all outcomes.
  The RLS-6 scale is an 11-point scale (from 0 = not present/completely satisfied to 10 = very severe/completely dissatisfied) to establish an individual severity profile at various day and night times (at bedtime; during the night; during the day when the patients are resting, or during the day when the patients are involved in daily activities).
Time Frame: From Baseline to end of Observation Period (3 months).
Population: Of the 564 subjects in the Full Analysis Set (FAS), 562 are included in this analysis.
  The FAS consists of all patients receiving treatment with Rotigotine at least once & for whom valid scores for item 2 & item 3 of the RLS-6 scale at baseline & at least one valid post baseline score for both item 2 & item 3 of the RLS-6 scale is documented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro®
Number analyzed (Participants) | 562
units on a scale
  Change from Baseline to End of Observation Period | -2.8 (3.2)
  Observed Value at Baseline Visit | 5.2 (2.8)

5. Secondary Outcome: Severity of Restless Legs Syndrome (RLS) at Daytime in Activity
Description: Severity of RLS at daytime in activity measured as change from baseline to end of observation period (Item 5 RLS-6 scale).
  The Last Observation Carried Forward (LOCF) method was utilized for all outcomes.
  The RLS-6 scale is an 11-point scale (from 0 = not present/completely satisfied to 10 = very severe/completely dissatisfied) to establish an individual severity profile at various day and night times (at bedtime; during the night; during the day when the patients are resting, or during the day when the patients are involved in daily activities).
Time Frame: From Baseline to end of Observation Period (3 months).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro®
Number analyzed (Participants) | 564
units on a scale
  Change from Baseline to End of Observation Period | -0.9 (2.3)
  Observed Value at Baseline Visit | 1.9 (2.4)

6. Secondary Outcome: Daytime Tiredness
Description: Daytime tiredness measured as change from baseline to end of observation period (Item 6 RLS-6 scale).
  The Last Observation Carried Forward (LOCF) method was utilized for all outcomes.
  The RLS-6 scale is an 11-point scale (from 0 = not present/completely satisfied to 10 = very severe/completely dissatisfied) to establish an individual severity profile at various day and night times (at bedtime; during the night; during the day when the patients are resting, or during the day when the patients are involved in daily activities).
Time Frame: From Baseline to end of Observation Period (3 months).
Population: Of the 564 subjects in the Full Analysis Set (FAS), 561 are included in this analysis.
  The FAS consists of all patients receiving treatment with Rotigotine at least once & for whom valid scores for item 2 & item 3 of the RLS-6 scale at baseline & at least one valid post baseline score for both item 2 & item 3 of the RLS-6 scale is documented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro®
Number analyzed (Participants) | 561
units on a scale
  Change from Baseline to End of Observation Period | -1.9 (3.2)
  Observed Value at Baseline Visit | 5.1 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected during the course of the trial, which was approximately 3 months per subject.
Description: Adverse Events refer to the Safety Set (SS). The Safety Set (SS) consisted of all patients included in this study receiving treatment with Neupro® at least once.
Arm/Group | Neupro®
Serious Adverse Events (participants affected / at risk) | 8/684
Other Adverse Events (participants affected / at risk) | 121/684
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neupro® (N=684)
Myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Radius fracture (Musculoskeletal and connective tissue disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Amaurosis fugax (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neupro® (N=684)
Nausea (Gastrointestinal disorders) | 39 (39)
Application site erythema (General disorders) | 8 (8)
Fatigue (General disorders) | 14 (14)
Headache (Nervous system disorders) | 19 (19)
Dizziness (Nervous system disorders) | 19 (19)
Sleep disorder (Psychiatric disorders) | 8 (8)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (23)
Rash (Skin and subcutaneous tissue disorders) | 15 (16)
Hypertension (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.